CLINICAL TRIAL: NCT07133659
Title: Exploring the Efficacy, Safety of a Modified Starting Dosage of Avatrombopag in Immune Throbocytopenia (ITP) - a Pilot Study
Acronym: Ava dosing
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Al-Mustansiriyah University (Other)
Responsible Party: Principal Investigator, Alaa Fadhil Alwan, consultant hematologist, Al-Mustansiriyah University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RGHC007
Record Dates: First submitted 2025-08-14; First posted 2025-08-21 (Actual); Last update posted 2025-08-21 (Actual); Status verified 2025-08

CONDITIONS: ITP - Immune Thrombocytopenia
Keywords: ITP; thrombocytopenia; Avatrombopag; thrombopoietin receptor agonist
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic; Thrombocytopenia | interventions — avatrombopag; Tablets

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Avatrombopag (Experimental): Description: Patients will start on avatrombopag 20 mg every other day for a week then the dose will be readjusted according to the platelet count.
  Interventions: Drug: Avatrombopag 20 mg Oral Tablet

INTERVENTIONS:
Drug: Avatrombopag 20 mg Oral Tablet — Description: Patients will start on avatrombopag 20 mg every other day for a week then the dose will be readjusted according to the platelet count.

SUMMARY:
This is a single-center, open label pilot trial where patients with primary ITP who require second line treatment will be offered avatrombopag at a reduced starting dose, adjusted thereafter according to the response and continued for up to 24 weeks. The study aims to acquire experience on use of avatrombopag and explore the efficacy and safety of lower starting dose of avatrombopag

DETAILED DESCRIPTION:
Avatrombopag is an oral thrombopoietin receptor agonist that is licensed for chronic ITP. Avatrombopag is administered at a starting dose of 20 mg daily. Overshooting of platelet count is a frequent problem that occurs in 20 to 40% of the patients after initiating avatrombopag as recommended. In this open label, single arm, pilot study, we will start avatrombopag at a reduced starting dose of 20 mg every other day. The dose will be adjusted thereafter according to the platelet response. The study consists of 3 phases: Dose adjustment phase, a maintenance phase, and dose tapering/disconsolation and follow-up phase. The study aims to acquire experience on use of avatrombopag and explore the efficacy and safety of lower starting avatrombopag-dose, and assess the rate of sustained response off-treatment. The duration of treatment with avatrombopag is 6 months.

The study is an investigator-initiated trial sponsored by Center for Transplantation and Blood Diseases. Medical City Complex, Baghdad Iraq.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female aged ≥18 years.
2. Diagnosis of primary ITP and having a platelet count of < 30 x109/L measured within two weeks prior to inclusion with failure to achieve response or relapse after at least one cycle of dexamethasone (20-40 mg daily for 4 days) or prednisone /prednisolone (1 mg/kg for at least two weeks). Shorter courses or lower doses are allowed if discontinued or modified due to side effects.
3. Clinical need for second (subsequent) line treatment with a platelet elevating therapy assessed by the physician in charge.
4. Signed and dated written informed consent.

Exclusion Criteria:

1. Previous treatment with TPO-RA.
2. Pregnancy or lactation.
3. Patients with active serious bleeding or at high risk of bleeding as judged by physician in charge.
4. Females of child-bearing potential refusing to follow effective contraceptive methods (as described in SmPC) during treatment with Avatrombopag.
5. Secondary ITP defined as ITP secondary to lymphoma or chronic lymphocytic leukemia; ITP secondary to the following autoimmune disorders Systemic Lupus Erythematosus or Antiphospholipid Syndrome; ITP secondary to Common Variable Immune Deficiency; ITP secondary to the following viral infections eg Human Immunodeficiency Virus.
6. Concomitant autoimmune hemolytic anemia, Evans syndrome.
7. Presence of any serious comorbidity where the condition may worsen the study drugs.
8. Presence of active malignancy unless deemed cured by adequate treatment. Participants with the following neoplastic conditions can be included:

   * Monoclonal gammopathy of undetermined significance (MGUS) or monoclonal B lymphocytosis of undetermined significance (MBUS)
   * Basal/squamous cell carcinoma of the skin
   * Carcinoma in situ of the cervix
   * Carcinoma in situ of the breast
   * Incidental histological finding of prostate cancer (TNM stage T1a or T1b)
9. Patients with history of poor compliance or history of alcohol/drug abuse or excessive alcohol beverage consumption that would interfere with the ability to comply with the study protocol, or current or past psychiatric disease that might interfere with the ability to comply with the study protocol or give informed consent.

   -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2025-06-08 (Actual); Primary Completion 2026-07-08 (Estimated); Study Completion 2027-07-08 (Estimated)

PRIMARY OUTCOMES:
Total Response Time | 20 weeks
  Median cumulative number of weeks with platelet count >50 x 109/L from time of Avatrombopag initiation to end of week 20. A period of 2 week will be deducted after IVIG and 4 weeks after dexamethasone.

SECONDARY OUTCOMES:
TTR | 20 weeks
  Time from initiation of dose to first platelet count > 50 x 109/L without any rescue therapy during the 2 weeks prior to the blood sampling.
Response by day 8 | 8 days
  Number of patients achieving platelet count > 50 x 109/L by day 8 without any rescue therapy during the 2 weeks prior to the blood sampling.
Rates of platelet overshoot. | 6 weeks
  Number of episode with platelet count > 200 and >400 x 109/L during the first 6 weeks after the initiation of avatrombopag.
Durable response rate. | 20 weeks
  Number of patients achieving 4 consecutive platelet counts > 50 x 109/L between weeks 12 and 20 including the last count, without the use of rescue therapy, corticosteroids or any platelet elevating agent after week 6.
The rates of treatment failure. | 20 weeks
  Occurrence of treatment failure is defined as:
  Discontinuation of Avatrombopag and switching to another platelet elevating agent between weeks 6 and 20 due to non-response or intolerance to Avatrombopag or administration of rescue therapy after week 6 and Thrombocytopenia (platelet count <30 x 109/L), high risk of bleeding or intolerance to avatrombopag.
Bleeding complications during the study. | 52 weeks
  Number and severity of WHO bleeding events.
The safety of treatment with Avatrombopag. | 52 weeks
  Occurrence and severity of treatment emergent adverse events. Occurrence and severity of adverse events of special interest including arterial and venous thrombosis and bone marrow fibrosis (bone marrow biopsy showing MF2 or higher).
The changes in HRQoL during the study. | 20 weeks
  Change in of SF-36 (v1) questionnaires from baseline to weeks 20.
The rates of Sustained Response Off-Treatment (SROT) at week 52. | 52 weeks
  Occurrence of SROT defined as:
  A platelet count > 30 x 109/L in all planned visits between the time of discontinuation of Avatrombopag and week 52 including week 52 and no administration of platelet elevating agent between weeks 20 and 52.

CONTACTS AND LOCATIONS:
Locations (1):
- hematology center / Medical City, Baghdad, Iraq

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Guillet S, Crickx E, Azzaoui I, Chappert P, Boutin E, Viallard JF, Riviere E, Gobert D, Galicier L, Malphettes M, Cheze S, Lefrere F, Audia S, Bonnotte B, Lambotte O, Noel N, Fain O, Moulis G, Hamidou M, Gerfaud-Valentin M, Marolleau JP, Terriou L, Martis N, Morin AS, Perlat A, Le Gallou T, Roy-Peaud F, Robbins A, Lega JC, Puyade M, Comont T, Limal N, Languille L, Zarrour A, Luka M, Menager M, Belmondo T, Hue S, Canoui-Poitrine F, Michel M, Godeau B, Mahevas M. Prolonged response after TPO-RA discontinuation in primary ITP: results of a prospective multicenter study. Blood. 2023 Jun 8;141(23):2867-2877. doi: 10.1182/blood.2022018665. PMID 36893453
- [Background] Pascual-Izquierdo C, Sanchez-Gonzalez B, Canaro-Hirnyk MI, Garcia-Donas G, Menor-Gomez M, Gil-Fernandez JJ, Monsalvo-Saornil S, de-Laiglesia A, Alvarez-Roman MT, Jarque-Ramos I, Llacer MJ, Pedrote-Amador B, Zafra-Torres D, Caparros-Miranda I, Ortuzar-Pasalodos A, Revilla-Calvo N, Bastida JM, Chica-Gullon E, Alvarellos M, Jimenez-Barcenas R, Bernat S, Martinez-Carballeira D, Lakhwani S, Lopez-Ansoar E, Moreno-Beltran ME, Lorenzo-Vizcaya A, Aguirre MA, Lasa-Eguialde M, Canet M, Gonzalez-Gascon-Y-Marin IT, Caballero-Navarro G, Cuesta A, Diaz-Lopez M, Arquero T, Moreno-Carbonell M, Mingot-Castellano ME; Spanish ITP Group (GEPTI) of the Spanish Society of Hematology and Hemotherapy (SEHH). Avatrombopag in immune thrombocytopenia: A real-world study of the Spanish ITP Group (GEPTI). Am J Hematol. 2024 Dec;99(12):2328-2339. doi: 10.1002/ajh.27498. Epub 2024 Oct 12. PMID 39394928
- [Background] Virk ZM, Leaf RK, Kuter DJ, Goodarzi K, Connell NT, Connors JM, Al-Samkari H. Avatrombopag for adults with early versus chronic immune thrombocytopenia. Am J Hematol. 2024 Feb;99(2):155-162. doi: 10.1002/ajh.27080. Epub 2023 Dec 8. PMID 38063420
- [Background] Yamaguchi H, Iino M, Kowata S, Yamamoto R, Yamanouchi J, Imamura Y, Kirito K, Yokoyama K, Ito T, Ishikawa T, Shiratsuchi M, Tomiyama Y, Kamiya H, Zhang J, Jamieson BD. A phase 3 study of the efficacy and safety of avatrombopag in Japanese adults with chronic immune thrombocytopenia. Int J Hematol. 2025 Oct;122(4):521-532. doi: 10.1007/s12185-025-04001-4. Epub 2025 May 20. PMID 40392465
- [Background] Tarantino MD, Bussel JB, Lee EJ, Jamieson BD. A phase 3, randomized, double-blind, active-controlled trial evaluating efficacy and safety of avatrombopag versus eltrombopag in ITP. Br J Haematol. 2023 Aug;202(4):897-899. doi: 10.1111/bjh.18908. Epub 2023 Jun 20. No abstract available. PMID 37339869
- [Background] Mei H, Zhou H, Hou M, Sun J, Zhang L, Luo J, Jiang Z, Ye X, Xu Y, Lu J, Wang H, Hui A, Zhou Y, Hu Y. Avatrombopag for adult chronic primary immune thrombocytopenia: a randomized phase 3 trial in China. Res Pract Thromb Haemost. 2023 Jul 26;7(6):102158. doi: 10.1016/j.rpth.2023.102158. eCollection 2023 Aug. PMID 37700877
- [Background] Jurczak W, Chojnowski K, Mayer J, Krawczyk K, Jamieson BD, Tian W, Allen LF. Phase 3 randomised study of avatrombopag, a novel thrombopoietin receptor agonist for the treatment of chronic immune thrombocytopenia. Br J Haematol. 2018 Nov;183(3):479-490. doi: 10.1111/bjh.15573. Epub 2018 Sep 7. PMID 30191972
- [Background] Matzdorff A, Alesci SR, Gebhart J, Holzhauer S, Hutter-Kronke ML, Kuhne T, Meyer O, Ostermann H, Pabinger I, Rummel M, Sachs UJ, Stauch T, Trautmann-Grill K, Wormann B. Expert Report on Immune Thrombocytopenia: Current Diagnostics and Treatment - Recommendations from an Expert Group from Austria, Germany, and Switzerland. Oncol Res Treat. 2023;46 Suppl 2:5-44. doi: 10.1159/000529662. Epub 2023 Feb 14. No abstract available. PMID 36787705
- [Background] Neunert C, Terrell DR, Arnold DM, Buchanan G, Cines DB, Cooper N, Cuker A, Despotovic JM, George JN, Grace RF, Kuhne T, Kuter DJ, Lim W, McCrae KR, Pruitt B, Shimanek H, Vesely SK. American Society of Hematology 2019 guidelines for immune thrombocytopenia. Blood Adv. 2019 Dec 10;3(23):3829-3866. doi: 10.1182/bloodadvances.2019000966. PMID 31794604
- [Background] Provan D, Arnold DM, Bussel JB, Chong BH, Cooper N, Gernsheimer T, Ghanima W, Godeau B, Gonzalez-Lopez TJ, Grainger J, Hou M, Kruse C, McDonald V, Michel M, Newland AC, Pavord S, Rodeghiero F, Scully M, Tomiyama Y, Wong RS, Zaja F, Kuter DJ. Updated international consensus report on the investigation and management of primary immune thrombocytopenia. Blood Adv. 2019 Nov 26;3(22):3780-3817. doi: 10.1182/bloodadvances.2019000812. PMID 31770441
- [Background] Rodeghiero F, Stasi R, Gernsheimer T, Michel M, Provan D, Arnold DM, Bussel JB, Cines DB, Chong BH, Cooper N, Godeau B, Lechner K, Mazzucconi MG, McMillan R, Sanz MA, Imbach P, Blanchette V, Kuhne T, Ruggeri M, George JN. Standardization of terminology, definitions and outcome criteria in immune thrombocytopenic purpura of adults and children: report from an international working group. Blood. 2009 Mar 12;113(11):2386-93. doi: 10.1182/blood-2008-07-162503. Epub 2008 Nov 12. PMID 19005182
- [Background] Ghanima W, Godeau B, Cines DB, Bussel JB. How I treat immune thrombocytopenia: the choice between splenectomy or a medical therapy as a second-line treatment. Blood. 2012 Aug 2;120(5):960-9. doi: 10.1182/blood-2011-12-309153. Epub 2012 Jun 26. PMID 22740443